CLINICAL TRIAL: NCT02314182
Title: GRECCAR 8 : Impact on Survival of the Primary Tumor Resection in Rectal Cancer With Unresectable Synchronous Metastasis a Randomized Multicenter Study
Brief Title: GRECCAR 8: Primary Tumor Resection in Rectal Cancer With Unresectable Metastasis
Acronym: GRECCAR8
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2014.847
Record Dates: First submitted 2014-11-12; First posted 2014-12-11 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Rectal Adenocarcinoma
Keywords: Rectal adenocarcinoma; unresectable; surgery; chemotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Drug Therapy; Oxaliplatin; Irinotecan; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A Primary tumor resection + chemotherapy (Experimental): PT resection + systemic chemotherapy +/- target therapy
  Interventions: Procedure: Primary tumor resection + chemotherapy
- B Oxaliplatin/irinotecan + capecitabine, 5-FUI ± bevacizumab (Other): Chemotherapy (+/- target therapy)
  Interventions: Drug: Oxaliplatin/irinotecan + capecitabine, 5-FUI ± bevacizumab

INTERVENTIONS:
Procedure: Primary tumor resection + chemotherapy — Step 1: Primary Tumor (PT) resection
  * Within 3 weeks after randomization
  * Immunonutrition given 7 days prior to PT resection
  * Mechanical bowel preparation performed before surgery according to the local practices
  * Performed by laparoscopy (recommended) or by laparotomy (at the investigator's discretion)
  Step 2: postoperative CT-scan
  * Must be performed within 4 weeks after surgery
  * CT-scan/MRI with the same criteria as pre-treatment evaluation
  Step 3: Chemotherapy +/- target therapy
  * Within 4 weeks after the surgery
  * Chemotherapy administered according to the usual scheme for the chosen protocol
  * All validated and/or registered perioperative rectal cancer treatments authorized
  * The duration of one treatment cycle depending on the type of treatment administered
  * Radiotherapy is allowed after randomization if indicated
  Arms: A Primary tumor resection + chemotherapy
Drug: Oxaliplatin/irinotecan + capecitabine, 5-FUI ± bevacizumab — Treatment will start within 3 weeks after randomization; Chemotherapy will be administered according to the regimen in the chosen protocol and validated by the MDOC of each center.
  If complications occur, emergency surgery can be performed according to the local practices of each investigator center.
  Radiotherapy is allowed after randomization if indicated (MDOC).
  Other Names: EGFR antibodies panitumumad and cetuxiamb in case of KRAS wild-type tumors.
  Arms: B Oxaliplatin/irinotecan + capecitabine, 5-FUI ± bevacizumab

SUMMARY:
A prospective, open, multicenter, randomized III trial with two arms:

* Arm A: Primary tumor resection , followed by chemotherapy
* Arm B: Chemotherapy alone. Compare overall 2-year survival rates in patients treated for resectable rectal adenocarcinoma with unresectable metastasis, treated either with the primary tumor resection with chemotherapy +/- target therapy, or with chemotherapy (+/- target therapy) alone.

ELIGIBILITY:
Inclusion Criteria:

* Non-complicated primary tumor (i.e. tumor without obstruction, bleeding, abscess or perforation requiring emergency surgery and/or contra-indicating first-line chemotherapy)
* Unresectable synchronous metastases
* ECOG performance status 0-1
* Rectal adenocarcinoma (<15 cm from the anal verge) with few or no symptoms and unresectable metastasis (assessed by the investigator) unsuitable for curative treatment
* No known unresectable primary tumor (with clear margin >1mm) on CT-scan and MRI
* No disease progression under chemotherapy (for at least 4 cycles);
* Assessment of KRAS status before randomization (wild type or mutated);
* Life expectancy without cancer >2 years
* White blood cell count ≥ 3 x 109/L, with neutrophils ≥ 1,5 x 109/L, platelet count ≥ 100 x 109/L, hemoglobin°≥ 9 g/dL (5,6 mmol/l)
* Total bilirubin ≤ 1.5 x ULN (upper limit of normal), ASAT and ALAT ≤ 2.5 x ULN, alkaline phosphatase°≤°1.5°x ULN, serum creatinine ≤ 1.5 x ULN;
* Age ≥ 18 years ≤ 75 years
* Patients with childbearing potential should use effective contraception during the study and up 6 months after the end of chemotherapy
* Covered by a Health System where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research;
* Signed written informed consent obtained prior to any study-specific screening procedures

Exclusion Criteria:

* Rectal tumor operated before inclusion
* Symptoms related to the rectal tumor requiring first intention rectal surgery (appreciated by investigator)
* Contra-indication for surgery
* Resectable metastases
* Complicated (obstruction, bleeding, abscess, perforation) primary tumor requiring emergency surgery and/or contra-indicating first line-chemotherapy
* Non-resectable primary tumor (with wild margin)
* Age > 75 years < 18 years
* ECOG performance status > 2
* Under nutrition (albumin < 30 g/l)
* Peritoneal carcinomatosis
* Disease progression under chemotherapy (RECIST 1.1 criteria)
* Known hypersensitivity reaction or specific contraindications to any of the components of study treatments
* Clinically relevant coronary artery disease or history of myocardial infarction in the last 12 months, or high risk of uncontrolled arrhythmia
* Pregnancy (absence to be confirmed by ß-hCG test) or breast-feeding;
* Previous malignancy in the last 5 years
* Medical, geographical, sociological, psychological or legal conditions that would prevent the patient from completing the study or signing the informed consent; in the investigator's opinion
* Any significant disease which, in the investigator's opinion, excludes the patient from the study
* Under an administrative or legal supervision.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-11-20 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02-27 (Actual)

PRIMARY OUTCOMES:
Overall survival | up to 2 years
  Overall survival, defined as the time interval between the date of randomization and the date of death, with a 24 months' follow-up, in both treatment arms.

SECONDARY OUTCOMES:
Progression free survival | up to 2 years
  Progression free survival will be assessed every 3 months during follow-up and will be estimated at 24 months.
Quality of life | Up to 2 years
  Quality of life will be assessed at the time of randomization and then every 3 months in both treatment arms. The EORTC QLQ-C30, QLQ-CR29 questionnaires will be used.
Toxicity of chemotherapy (Common Toxicity Criteria for Adverse Events (NCI-CTC-AE V4.0) | Up to 2 years
  Chemotherapy toxicity will be graded according to the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTC-AE V4.0) in both treatment arms
Response of the metastatic disease to systemic chemotherapy (RECIST 1.1 criteria) | up to2 years
  The response rate of the metastatic disease will be evaluated in both treatment arms by CT scan and analyzed using the RECIST 1.1 criteria
Time to disease progression | up to 2 years
  Time to disease progression is defined as the lapse of time between the date of randomization and the first date of progression (clinical or imaging) of the metastatic disease in both treatment arms, or of the primary rectal tumor in the chemotherapy arm (Arm B)
Post-operative morbidity | within 30 days after surgical intervention
  The evaluation of post-operative morbidity and mortality will be assessed in the primary tumor resection arm (Arm A) and in the chemotherapy arm (Arm B) for patients who require emergency surgery. The post-operative complications will be evaluated according to the Clavien-Dindo Classification of Surgical Complication and graded 0 to V.

CONTACTS AND LOCATIONS:
Overall Officials: Eddy COTTE, Principal Investigator — Service de Chirurgie Générale et Digestive, Centre hospitalier Lyon Sud, HCL
Locations (3):
- France (3):
  - Service de Chirurgie Générale et Digestive, Centre hospitalier Lyon Sud, HCL, Pierre-Bénite, France
  - Service d'Oncologie Médicale, Clinique du Cap-d'Or, La Seyne-sur-Mer
  - Service de Chirurgie Générale et Digestive, CHRU Claude Huriez, Lille

REFERENCES:
- [Result] Cotte E, Villeneuve L, Passot G, Boschetti G, Bin-Dorel S, Francois Y, Glehen O; French Research Group of Rectal Cancer Surgery (GRECCAR). GRECCAR 8: impact on survival of the primary tumor resection in rectal cancer with unresectable synchronous metastasis: a randomized multicentre study. BMC Cancer. 2015 Feb 12;15:47. doi: 10.1186/s12885-015-1060-0. PMID 25849254